CLINICAL TRIAL: NCT05955820
Title: Effect of a Selected Suspension System Exercise Program on Patients With Subacromial Impingement Syndrome
Brief Title: Suspension System on Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Mumdouh Yousef, PROF.DR.Enass Fawzy Youssif, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Impingement syndrome new EX
Record Dates: First submitted 2023-07-08; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Impingement Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional exercises for impingement syndrome (Experimental): Four exercises (prone extension, side-lying external rotation, side-lying forward flexion, prone horizontal abduction with external rotation) will be performed for three sets of 10 repetitions
  Interventions: Device: Dumbbells
- Suspension system exercises for impingement syndrome (Experimental): Four exercises (Kneeling shoulder extension, Supine/ standing / kneeling row, sitting press up, kneeling push up) will be performed for 3-6 sets of 10 repetitions
  Interventions: Device: Suspension system

INTERVENTIONS:
Device: Suspension system — Participants will be tested by four exercises designed for impingement syndrome using the suspension system
  Other Names: Neurac system
  Arms: Suspension system exercises for impingement syndrome
Device: Dumbbells — Participants will be tested by four exercises designed for impingement syndrome using Dumbbells
  Arms: Conventional exercises for impingement syndrome

SUMMARY:
To investigate the effect of shoulder exercise using a selected suspension system exercise program on pain, disability, functional performance and proprioception in patients with subacromial impingement syndrome.

DETAILED DESCRIPTION:
Two groups were assigned to this study, the first one received four conventional exercises that designed for shoulder impingement syndrome, the second group received the same four conventional exercises plus four selected suspension system exercises.

The sessions were conducted three times per week fir four weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Fifty-eight subjects with SIS (more than three months).
2. Their age ranges from 20-45 years old
3. Level of pain (at least 2/10 on VAS)
4. Body mass index (BMI) between 18-25
5. Subjects must show positive results in at least two of the following tests: Neer's impingement test, Hawkins-Kennedy test, supraspinatus (empty can) test, apprehension and relocation test.

Exclusion Criteria:

The subjects will be excluded if they had:

1. Received physiotherapy at last 3 months.
2. Received corticosteroids injection in subacromial space at last 3 months.
3. Received anti-inflammatory medications.
4. Have a fracture or dislocation in shoulder, neck and thoracic regions.
5. Have an acute rotator cuff tear.
6. Have tumor or malignancy in shoulder region.
7. Have neurologic problems in shoulder, neck and thoracic regions.
8. Have cooperation difficulties due to cognitive disorders.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
Improvement in active shoulder ROM | Baseline
  Proprioception will be tested by using inclinometer to determine patient's active shoulder range of motion for internal and external rotation, flexion, and extension
Improvement in functional performance | Baseline
  Assessment of function using SPADI subscale which contains 13 items that assess two domains; a 5-item subscale that measures pain and 8-item subscale that measures disability. In addition, Several non-specific strength/power tests may assist in determining the level of functional performance of the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university faculty of physical therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen L, Chen J, Peng Q, Chen J, Zou Y, Liu G. Effect of Sling Exercise Training on Balance in Patients with Stroke: A Meta-Analysis. PLoS One. 2016 Oct 11;11(10):e0163351. doi: 10.1371/journal.pone.0163351. eCollection 2016. PMID 27727288